CLINICAL TRIAL: NCT03787524
Title: Prediction of Functional Health Status and Aspiration Using Multiple Dysphagia Scales Over 6 Months After Acute Stroke: Prospective, Observational, Parallel Group, Case-control Trial
Brief Title: Prediction of Functional Health Status and Aspiration Using Multiple Dysphagia Scales Over 6 Months After Acute Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Associate Professor, Ulsan University Hospital
Other Study IDs: chhwang12
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Acute Stroke; Dysphagia
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysphagia group: Acute stroke patients who will be diagnosed dysphagia according to VFSS results.
- No dysphagia group: Acute stroke patient who showed no dysphagia according to VFSS results.

SUMMARY:
In order to discover dysphagia scales, which shows meaningful predictability of aspiration and functional health status in patients with acute stroke, authors plan to find out more predictable indicators than existing penetration-aspiration scale (PAS) to validate their predictions and their internal and external validity over 6 months following stroke .

DETAILED DESCRIPTION:
To determine the dysphagia scale with significant predictions of aspiration and functional health status in patients with acute stroke, video-fluoroscopic swallowing study (VFSS) will be performed to the patients who will be referred for VFSS among stroke patients who would be diagnosed by Brain MRI / CT. When any type of dysphagia is found, participant will be assigned to the test group (DYS), and when no dysphagia is found, they will be assigned to the control group (NOD).

Numerous kinds of assessment will be conducted before and after VFSS, before discharge, and 3, 6, and 9 months after the stroke onset.

ELIGIBILITY:
Inclusion Criteria:

* brain MRI / CT-based stroke patients who were referred for VFSS

Exclusion Criteria:

* In case of a history of dysphagia
* Unstable patient in neurology
* 2 or higher of NIHSS 1a (level of consciousness)
* Patients with other neurological diseases
* Patients with decompression skull resection
* Refusal of participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the raw data of BMI by Batsis et al's report in 2017 (mean value of two groups: 28.5 and 27.6, mean SD of two groups: 1.0), authors calculated total numbers of subjects, based on the Kang method using G power 3.1. Assuming the between factors analysis using the F-test of MANOVA, effect size 0.45, α value ≤0.05, power 0.8, number of groups 2, and number of repeated measures 4 were inputted. Supposed that the dropout rate was 20%, 34 patients in each group were finally calculated.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of Body mass index (Kg/m2) | 1 day before and 1 day, 3 weeks after the VFSS, 3 month, 6 months and 9 months after the stroke onset
  Body mass index (Kg/m2)

SECONDARY OUTCOMES:
Check the Penetration/aspiration on PAS | 1 day after the VFSS, 3 month, 6 months and 9 months after the stroke onset
  Penetration/aspiration on PAS (DYS)

OTHER OUTCOMES:
Change of Grasping force (kg) | 1 day before and 1 day, 3 weeks after the VFSS, 3 month, 6 months and 9 months after the stroke onset
  Grasping force (kg)
Change of Korean-modified Barthel index | 1 day before and 1 day, 3 weeks after the VFSS, 3 month, 6 months and 9 months after the stroke onset
  Korean-modified Barthel index: 0-100: the higher, the better
Change of Swallowing-Quality of Life | 1 day before and 1 day, 3 weeks after the VFSS, 3 month, 6 months and 9 months after the stroke onset
  Swallowing-Quality of Life: 1-44: the higher, the worse
Check the Aspiration pneumonia | 1 day, 3 weeks after the VFSS, 3 month, 6 months and 9 months after the stroke onset
  number of participants diagnosed aspiration pneumonia
Change of Eating Assessment Tool | 1 day, 3 weeks after the VFSS, 3 month, 6 months and 9 months after the stroke onset
  Eating Assessment Tool
change of Video-fluoroscopic Dysphagia Scale | 1 day after the VFSS
  Video-fluoroscopic Dysphagia Scale (VDS); 0-100; the higher, the worse
Modified Barium Swallowing Study Impairment Profile | 1 day after the VFSS
  Modified Barium Swallowing Study Impairment Profile (MBSImP); 0-62; the higher, the worse
Dynamic Imaging Grade of Swallowing Toxicity | 1 day after the VFSS
  Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) Scale; 0-4; the higher, the worse
Dysphagia Item of Common Terminology Criteria for Adverse Events | 1 day after the VFSS
  Dysphagia-related Item score, based on the Common Terminology Criteria for Adverse Events (CTCAE); 0-4; the higher, the worse
American Speech-Language Hearing Association National Outcomes Measurements System Swallowing Scale | 1 day after the VFSS
  American Speech-Language Hearing Association National Outcomes;Measurements System Swallowing Scale (ASHA NOMS); 1-7; the higher, the better
Confirmation of death | 3 month, 6 months and 9 months after the stroke onset
  number of participant of death confirmation

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D., Ph.D., Study Director — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea